CLINICAL TRIAL: NCT03189771
Title: Effect of Occlusal Reduction on Post-operative Pain in Patients With Irreversible Pulpitis and Symptomatic Apical Periodontitis Treated in a Single-visit: A Randomized Clinical Trial
Brief Title: Effect of Occlusal Reduction on Post-operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fadwa sheesh, Bachelor degree of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: evidence comittee
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Evaluate Occlusal Reduction on Post-operative Pain; Teeth With Symptomatic Irreversible Pulpitis; Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusal surface reduction (Experimental): occlusal surface reduction after single visit root canal treatment
  Interventions: Procedure: occlusal surface reduction
- no occlusal surface reduction (Placebo Comparator): No occlusal surface reduction after single visit root canal treatment
  Interventions: Procedure: occlusal surface reduction

INTERVENTIONS:
Procedure: occlusal surface reduction — occlusal surface reduction after single visit root canal treatment

SUMMARY:
effect of occlusal reduction on post-operative pain is evaluated after single visit root canal treatment in upper and lower molar teeth in patients with sypmtomatic irreversible pulpitis and apical periondontis

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between 20-50 years with no sex predilection.
2. Medically free patients.
3. Patients suffering from symptomatic irreversible pulpitis with symptomatic apical periodontitis in maxillary and mandibular molars with:

   * Preoperative pain.
   * Vital pulp.
   * Sensitivity to percussion.
   * Occlusal contact with the opposing teeth.
   * Normal periapical radiographic appearance or slight widening in the periodontal membrane space.

Exclusion Criteria:

1. Pregnant females.
2. Patients having a significant systemic disorder.
3. Patients who had administered analgesics or antibiotics during the last 12 hours preoperatively.
4. Patients having bruxism or clenching.
5. Teeth having :

   * No occlusal contact.
   * No sensitivity to percussion.
   * Association with swelling or fistulous tract.
   * Acute or chronic peri-apical abscess.
   * Greater than grade I mobility.
   * Pocket depth greater than 5mm.
   * No possible restorability.
   * Previous endodontic treatment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-06-27 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
pre-operative pain before single visit root canal treatment by NRS (numerical rating scale) | Baseline
  Primary outcome will be assessed by NRS (numerical rating scale), the unit of measurement is categorical.The scale is from (0-10) (1-3) Mild pain (4-6) Moderate pain (7-10) Severe pain
post-operative pain after single visit root canal treatment by NRS (numerical rating scale) | after treatment by 6 hours
  Primary outcome will be assessed by NRS (numerical rating scale), the unit of measurement is categorical.The scale is from (0-10) (1-3) Mild pain (4-6) Moderate pain (7-10) Severe pain
post-operative pain after single visit root canal treatment by NRS (numerical rating scale) | after treatment by 12 hours
  Primary outcome will be assessed by NRS (numerical rating scale), the unit of measurement is categorical.The scale is from (0-10) (1-3) Mild pain (4-6) Moderate pain (7-10) Severe pain
post-operative pain after single visit root canal treatment by NRS (numerical rating scale) | after treatment by 24 hours
  Primary outcome will be assessed by NRS (numerical rating scale), the unit of measurement is categorical.The scale is from (0-10) (1-3) Mild pain (4-6) Moderate pain (7-10) Severe pain
post-operative pain after single visit root canal treatment by NRS (numerical rating scale) | after treatment by 48 hours
  Primary outcome will be assessed by NRS (numerical rating scale), the unit of measurement is categorical.The scale is from (0-10) (1-3) Mild pain (4-6) Moderate pain (7-10) Severe pain

IPD SHARING:
Plan to Share IPD: No